CLINICAL TRIAL: NCT06486194
Title: Analytical Validation and Clinical Testing of the Preemie System for Analysis and Calculation of Targeted Fortification of Mother's Breast Milk for Preterm Infants
Brief Title: Preemie Milk Analyser Validation Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: Tellspec Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CHI1219
Record Dates: First submitted 2024-06-10; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Pre-Term; Breast Milk Expression; Nutrition Disorder, Infant
MeSH Terms: conditions — Premature Birth; Breast Milk Expression; Infant Nutrition Disorders

STUDY DESIGN:
Intervention Model Description: Phase 1: Validation of the Preemie sensor, encompassing 2 different analytical studies for assessing the accuracy (1) and the precision/reproducibility (2) of the system
  Phase 2: Open label randomised controlled trial to test use of Preemie ecosystem in clinical practice for the delivery of targeted individualised breast milk fortification
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Targeted breast milk fortification using preemie device (Experimental): Mother's breast milk (MBM) or Donor Breast Milk (DBM) for use in a day's milk feeds will be measured using the Preemie sensor every 2-3 days, results recorded, and the amounts of breast milk fortifier (BMF), protein supplement, carbohydrate supplement and fat supplements needed to be added in order for that sample of milk to meet current 2022 European Society of Pediatric Gastroenterology, Hepatology and Nutrition (ESPGHAN) enteral nutrient intake recommendations calculated by the Preemie Sensor NutriNTrack software. Feeds will be made up in batches of 24hrs worth of feeds each day based on these calculations and the resulting supplement amounts used for the next 2-3 days until another sample of MBM is analysed, in line with previous work by Rochow et al
  Interventions: Device: Targeted breast milk fortification using preemie device; Dietary Supplement: Standard Breast milk fortification
- Standard Fortification (Active Comparator): Mother's breast milk (MBM) or Donor Breast Milk (DBM) for use in a day's milk feeds will be measured using the Preemie sensor every 2-3 days and results recorded. Breast milk will then be fortified in the standard way according to the manufacturer's recommendations, which assume a standard macronutrient content of the milk.
  Interventions: Dietary Supplement: Standard Breast milk fortification

INTERVENTIONS:
Device: Targeted breast milk fortification using preemie device — Mother's breast milk will have additional macronutrient added to it based on analysis with the Preemie device, to ensure it meets current European recommendations for nutrient intakes for preterm infants
  Arms: Targeted breast milk fortification using preemie device
Dietary Supplement: Standard Breast milk fortification — Standard multicomponent breast milk fortifier will be added to mother milk as per usual practice for preterm infants

SUMMARY:
This study aims to test and validate the Preemie Ecosystem- a new device and associated software package for measuring the nutrient (fat, protein and carbohydrate) content of the breast milk of the mothers of premature babies. This is potentially useful, as premature babies have higher nutritional requirements than babies born at term near their due date. At the moment, a nutritional supplement called breast milk fortifier is added to breast milk in standard amounts to improve its nutritional content and help premature babies grow. However, we know that each mother's breast milk is different, and varies from day to day, so each mother's milk may require more or less of such supplements in order to meet European recommendations for the nutrient intake.

The aim of this study is to first test and validate the accuracy of the Preemie device for measuring the nutritional content of mother's breast milk, using milk donated to the local donor milk bank and from mothers of babies currently on the neonatal unit. Next, once this is complete, the aim is to demonstrate it is feasible to use the Preemie device to enable fortification of mother's milk on an individualised basis for a small group of premature babies. The growth and nutrient intakes of these babies will be compared to another group who are cared for using the standard fortification approach.

The results of this study will be used to gain "Conformité Européenne" (CE) certification of the Preemie device and software.

DETAILED DESCRIPTION:
This is a single centre study taking place in a neonatal intensive care unit which is a regional referral centre for neonatal surgery and other tertiary specialities. The centre has well established policies for nutritional care, inducing the routine use of breast milk fortifier, and a track record in research into the nutrition and growth of preterm infants. It will have 2 phases:

Phase 1: Validation of the Preemie sensor, encompassing 2 different analytical studies for assessing the accuracy (1) and the precision/reproducibility (2) of the system

Phase 2: Open label randomised controlled trial to test use of Preemie ecosystem in clinical practice for the delivery of targeted individualised breast milk fortification

The methods used in each phase are as follows:

PHASE 1: Validation of Preemie Sensor Part A - Mothers currently expressing breast milk and meeting the inclusion criteria will be approached to take part in the study. They will be asked to provide 120ml of their breast milk which will be divided into a 20ml sample for use with the Preemie system and a 100ml sample for formal laboratory testing. The 20ml will be divided into ten smaller 2ml samples, and these will have their nutrient content (energy, fat, carbohydrate/sugar and protein) measured each day (in triplicate) using the Preemie sensor over a five day period and results recorded. The 100ml sample will be sent away to an independent third-party external laboratory to have its nutrient content (energy, fat, carbohydrate and protein) measured using standardised laboratory methods and results returned back to the study team. The results from the 2 systems will then be compared and the Preemie sensor assessed for accuracy.

Part B - 5 mothers currently expressing milk and donating to Southampton Milk bank will be approached to take part in the study and asked to provide 170ml of their milk which will be divided into a 100ml sample for formal laboratory testing (see above). For reproducibility tests, the 5 milk samples (30 aliquots of 2 mL per sample for running the test, and 5 aliquots serving as back-up, for a total of 70 ml per sample) will be analysed in 3 different rooms, by 3 different operators, using independent Preemie units, over the 5-day precision study. The Preemie precision/reproducibility will be then assessed by measuring the standard deviation between day, within run, between run, and in total, at each site, for each analyte.

For purposes of this phase of the study a "human breast milk sample" is one provided by a mother from a single expression. A mother may provide more than one sample if her milk supply allows this (see inclusion criteria) but samples should be at least 3 weeks apart. Purposive sampling will be used to ensure that the source of the samples is spread equally across the following 3 groups:

* Mothers of preterm infants born before 37 weeks gestation
* Mothers of term infants less than 8 weeks old
* Mothers of term infants more than 8 weeks old

PHASE 2: Open label randomised controlled trial to test use of Preemie ecosystem in clinical practice for the delivery of targeted individualised breast milk fortification This phase will see if it is possible to recruit to a trial and deliver targeted fortification of breast milk for infants on the Neonatal Intensive Care Unit (NICU) to improve their growth and metabolism.

30 preterm infants will be recruited and randomised (chosen at random using a computer) to receive either targeted fortification or standard fortification. In the targeted fortification group, the nutritional content (energy, fat, carbohydrate and protein) of mothers breast milk (MBM) or Donor Breast Milk (DBM) for use in a days milk feeds will be measured using the Preemie sensor every 2-3 days, and the amounts of breast milk fortifier (BMF), Protein supplements, carbohydrate supplements and fat supplements needed to be added in order for that sample of milk to meet current 2022 European recommendations nutritional intake for preterm infants calculated by the Preemie Sensor NutriNTrack software. Feeds will be made up in batches of 24hrs worth of feeds each day based on these calculations and the resulting supplement amounts used for the next 2-3 days until another sample of MBM is analysed. This approach is in line with the research of other groups who have demonstrated this approach to be safe (using a different milk analyser). In the Standard fortification group Mother's breast milk (MBM) or Donor Breast Milk (DBM) for use in a days milk feeds will be measured using the Preemie sensor every 2-3 days and results recorded. MBM or DBM will then be fortified in the standard way according to the manufacturer's recommendations, which assume a standard macronutrient content of the milk The allocated fortification approach (targeted or standardised) will be continued until the infant no longer requires fortification (eg moves onto formula milk) or reaches 34 weeks (when they would begin to have some breast feeds), is transferred to another hospital, or discharged home At the end of the study the two sets of infants will be compared in terms of nutrient intakes and growth.

Staff involved in delivering the Targeted Fortification will also be asked to provide feedback on the ease of use of the Preemie Ecosystem through semi-structured interviews and focus groups. Staff may also be observed by research staff using the machine in order to understand any issues and improve ease of use and user experience.

ELIGIBILITY:
Inclusion criteria Phase 1A For University Hospital Southampton (UHS) milk bank donors

* Approved as a donor for the UHS milk bank through the usual process
* Be providing milk to UHS donor milk bank For mothers of infant inpatients
* Have an infant who is currently an inpatient in the neonatal unit, paediatric wards, paediatric cardiac ward, or paediatric intensive care unit
* Be providing breastmilk for their preterm or term born infant
* Have sufficient breast milk available such that providing 120ml breast milk for the study does not impact on the needs of their infant.

Inclusion criteria Phase 1B

* Approved as a donor for the UHS milk bank through the usual process
* Be providing milk to UHS donor milk bank

Exclusion criteria Phase 1A and 1B For mothers of infant inpatients

- Mothers whose infants are inpatients and where there is a concern about adequacy of maternal milk supply to feed their infant

Inclusion Criteria Phase 2

* Birth weight ≥1kg and <1.8 kg (so meet the ESPGHAN criteria for breast milk fortification)
* Be taking fully fortified enteral breast milk feeds (≥150 ml/kg/day of mothers or donor breast milk containing breast milk fortifier as per the manufacturer's instructions)
* Tolerating fully fortified breast milk feeds≥150 ml/kg/day for 48 hours
* No longer on parenteral nutrition.

Exclusion Criteria Phase 2

* Infants where there is a concern about mother's supply of breast milk being insufficient to meet demands (where donor milk is not being used to make up any shortfall);
* Known congenital metabolic disorder;
* Infant formula fed;
* Bilateral grade III or IV intraventricular haemorrhage;
* Any infant who has had gastrointestinal tract surgery;
* Refusal of consent;
* Refusal for the use of breast milk fortifier
* Birthweight <1 kg

Ages: 0 Days to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Accuracy of the Preemie system against reference laboratory International Standards Organization (ISO) methods. | 6 months
  Establish accuracy of the Preemie system in measuring the macronutrient content of human milk (fat in g/L, fatty acids in g/L, protein in g/L, carbohydrate in g/L, and energy in g/L) carried out using the Preemie system and determining the bias against the same measurements performed through validated reference laboratory methods; Accuracy study of the Preemie system by paired testing of at least 100 human breast milk samples using both the Preemie system and reference laboratory ISO methods As per the Clinical and Laboratory Standards (CLSI) reference standard EP09c, Measurement Procedure Comparison and Bias Estimation Using Patient Samples - 3rd Edition, 2018, the accuracy of the Preemie system compared to the reference laboratory will be assessed through regression analysis, method comparison (R2, slope, intercept calculations), and bias estimations at low, medium, and high levels of each analyte.
Phase 1: Precision of the Preemie system against reference laboratory ISO methods. | 6 months
  Establish precision/reproducibility of the Preemie sensor by assessing the standard deviation of measures of the macronutrient content of human breast milk (protein in g/L, Fat in g/L, carbohydrate in g/l) related to measurements collected by different operators and units Precision/reproducibility study of the Preemie system by paired testing of at least 5 human milk samples.
  As per the CLSI reference standard EP05-A3, Evaluation of Precision of Quantitative Measurement Procedures; Approved Guideline - 3rd Edition, 2014, the Preemie system precision/reproducibility will be assessed by measuring the standard deviation between day, within run, between run, and in total, at each site, for each analyte.
Phase 2: Feasibility of recruiting infants to a study using Preemie system and associated NutriNTrack software to provide targeted individualised breast milk fortification in line with European recommendations. | 1 year
  Measure ability to recruit infants to study (recruitment success rates given as the percentage of parents giving consent of the total number approached)
Phase 2: Feasibility of using Preemie system and associated NutriNTrack software to provide targeted individualised breast milk fortification in line with European recommendations. | 1 year
  Measure ability to deliver intervention successfully (intervention compliance given as a percentage of infants randomised to targeted individualised breast milk fortification who received the intervention as intended)

SECONDARY OUTCOMES:
Phase 2: Enteral macronutrient intakes | 36 weeks corrected gestational age
  Compare enteral macronutrient (energy, carbohydrate, protein and fat) intake in g/kg/day as measured by the Preemie system in treated groups compared to non-treated groups during duration of treatment period.
Phase 2: Enteral trace element intakes | 36 weeks corrected gestational age
  Compare enteral trace elements (zinc, selenium and copper) intakes in mcg/kg/day as calculated based on measured milk intake in treated groups compared to non-treated groups during duration of treatment period.
Phase 2: Enteral fat-soluble vitamin intakes | 36 weeks corrected gestational age
  Compare fat-soluble vitamin (A, D, E and K) intake in units/kg/day as calculated based on measured milk intake in treated groups compared to non-treated groups during duration of treatment period.
Phase 2: Enteral wate-soluble vitamin intakes | 36 weeks corrected gestational age
  Compare water-soluble vitamin (C and B vitamins) intake in mcg/kg/day as calculated based on measured milk intake in treated groups compared to non-treated groups during duration of treatment period.
Phase 2: Enteral electrolyte intakes | 36 weeks corrected gestational age
  Compare enteral electrolytes (sodium, potassium, magnesium, phosphate, calcium) intake in mmol/kg/day as calculated based on measured milk intake in treated groups compared to non-treated groups during duration of treatment period.
Phase 2: Feed intolerance | 36 weeks corrected gestational age
  Establish days of feed intolerance in each group (defined as number of days enteral feed was withheld for =>12 hours due to concerns about nasogastric aspirate colour or volume, vomiting, abdominal distension, stooling or vomiting) as a proportion of the total number of days on which standard or targeted individualised breast milk fortification was included in the feed and compare between groups
Phase 2: Neonatal morbidities | 36 weeks corrected gestational age
  Compare rates of major neonatal morbidity between groups, consisting of necrotising enterocolitis (NEC), bronchopulmonary dysplasia (BPD, defined as requirement for oxygen beyond 36 weeks corrected gestational age), and culture positive sepsis.
Phase 2: Ease of use of Preemie device | 1 year (end of study)
  Obtain feedback from clinical staff on the process of targeted fortification using the Preemie sensor and software, including ease of use, time taken and complexity, clinical relevance, etc
Phase 2: Weight Gain | 36 weeks corrected gestational age
  Change in standard deviation score for weight (in kg) between birth and 36 weeks corrected gestational age
Phase 2: Head Growth | 36 weeks corrected gestational age
  Change in standard deviation score for head circumference (in cm) between birth and 36 weeks corrected gestational age
Phase 2: Length Growth | 36 weeks corrected gestational age
  Change in standard deviation score for length (in cm) between birth and 36 weeks corrected gestational age
Phase 2: Urea as a serum marker of nutritional status | 36 weeks corrected gestational age
  Compare mean serum urea (mmol/L) each week of the study between groups
Phase 2: Albumin as a serum marker of nutritional status | 36 weeks corrected gestational age
  Compare mean serum albumin urea (g/L) each week of the study between groups
Phase 2: Alkaline Phosphatase (ALP) as a serum marker of nutritional status | 36 weeks corrected gestational age
  Compare mean serum alkaline phosphatase (U/L) each week of the study between groups

CONTACTS AND LOCATIONS:
Overall Officials: Mark J Johnson, PhD, Principal Investigator — University Hospital Southampton NHS Foundation Trust
Locations (1):
- University Hospital Southampton NHS Foundation Trust, Southampton, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No